CLINICAL TRIAL: NCT03614143
Title: Biomarker Identification for aGVHD After Allogeneic Stem Cell Transplantation: a Multiple Center Study
Brief Title: Biomarker Study for Prediction of aGVHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Deputy director, department of hematology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHTG-001
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: aGVHD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective study in patients receiving allogeneic stem cell transplantation. The blood samples on Day-14, -7, 0 and every 7 days until D100 were collected together with clinical data. In the final analysis, cytokines and biomarkers analysis will be carried out and compared between patients in No aGVHD and grade II-IV aGVHD.

DETAILED DESCRIPTION:
This is a prospective study, observation study in patients receiving allogeneic stem cell transplantation in 4 BMT centers in Shanghai. The blood samples (on Day-14, -7, 0 and every 7 days until D100) and clinical data will be collected. In the final analysis, a panel of cytokines and biomarkers analysis of serial blood samples will be carried out and compared between patients with no aGVHD and grade II-IV aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing allogeneic stem cel transplantation
* with informed consent
* patients survived without aGVHD or relapse and patients with development of grade II-IV aGVHD

Exclusion Criteria:

* patients with blood sample and clinical data not available

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients received allogeneic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
incidence of grade II-IV aGVHD | 100 days after allogeneic stem cell tansplantation
  clinical diagnosis and grade of aGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No